CLINICAL TRIAL: NCT01870362
Title: Improvement of Periodontal Health and Reduction in Periodontal Plaque Micro-flora Using a Probiotic Lozenge in Patients With Chronic Periodontitis
Brief Title: Efficacy of a Probiotic Lozenge (Inersan) in Patients With Chronic Periodontitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CD Pharma India Pvt. Ltd. (Industry)
Collaborators: Mahatma Gandhi Post-Graduate Institute of Dental Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: prob-gracetpaul_01
Record Dates: First submitted 2013-06-03; First posted 2013-06-06 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Inersan) Arm (Experimental): Inersan Lozenges (2 Lozenges bid). Each probiotic lozenge contains not less than 1 billion CFU of L. brevis CD2
  Interventions: Drug: Probiotic (Inersan)
- Placebo Arm (Placebo Comparator): Placebo Lozenges (2 lozenges bid). Placebo lozenge contains only excipients (without probiotic).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Probiotic (Inersan)
  Other Names: Inersan contains not less than 1 billion CFU of Lactobacillus brevis CD2
  Arms: Probiotic (Inersan) Arm
Drug: Placebo
  Other Names: Placebo contains all excipients except the active constituent (Lactobacillus brevis CD2)
  Arms: Placebo Arm

SUMMARY:
Periodontal disease is a major cause of tooth loss in humans and is one of the most prevalent diseases associated with bone loss. Following bacterial colonization, the gingiva becomes inflamed leading, in some cases, to the destruction of the alveolar bone. Periodontitis has two distinct but interconnected etiologic components, periodontopathic bacteria and host-mediated connective tissue-destructive responses to the causative bacteria and their metabolic products.

A few studies have revealed that probiotic Lactobacillus strains were useful in reducing gingival inflammation and the number of black-pigmented rods, including Porphyromonas gingivalis (Pg), in the saliva and sub-gingival plaque. Concerning periodontal conditions, its shown that application of beneficial bacteria, as an adjunct to scaling and root planing (SRP), can inhibit re-colonization of pathogens in periodontal pockets and reduce bleeding on probing.

The aim of the present study is to evaluate the improvement of periodontal health with probiotic (Inersan) lozenges, used as an adjunct to scaling and root planing [SRP].

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes
* Patients in the age group of 25-60 years
* Subjects with mild to moderate chronic periodontitis, as defined by probing pocket depths 5-7mm in > 30 % of the probing sites
* The subjects should have at least 16 remaining natural teeth (minimum of at least 4 teeth per quadrant)
* Subjects in good general health

Exclusion Criteria:

* No antibiotic therapy in the past 2 months
* Medically compromised patients
* Subjects who are pregnant/ lactating
* Smokers and/or alcoholics.
* Those who had undergone any dental surgical or non-surgical therapy within 6 months prior to the start of the study.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2013-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Improvement in periodontal indices | 6 weeks, 12 weeks
  Improvement in Periodontal indices, namely, plaque index [PI], Gingival index [GI], Gingival bleeding index [GBI], probing pocket depth [PPD] and clinical attachment levels [CAL] in both groups

SECONDARY OUTCOMES:
Microbiological indices | 6 weeks, 12 weeks
  Changes in pathogen (Aggregatibacter actinomycetemcomitans (Aa), Porphyromonas gingivalis (Pg), and Prevotella intermedia) levels

CONTACTS AND LOCATIONS:
Overall Officials: Grace T Paul, MBBS, MDS, Principal Investigator — Mahatma Gandhi Post- Graduate Institute of Dental Sciences, Pondicherry
Locations (1):
- Mahatma Gandhi Post Graduate Institute of Dental Sciences (MGPGI), Puducherry, Puducherry, India